CLINICAL TRIAL: NCT06131983
Title: A Phase1/2a Dose-Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ARO-DUX4 in Adult Patients and Adolescent Patients With Facioscapulohumeral Muscular Dystrophy Type 1
Brief Title: Study of ARO-DUX4 in Adult and Adolescent Patients With Facioscapulohumeral Muscular Dystrophy Type 1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARODUX4-1001
Record Dates: First submitted 2023-11-08; First posted 2023-11-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Facio-Scapulo-Humeral Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-DUX4 (Experimental): ARO-DUX4 for Injection
  Interventions: Drug: ARO-DUX4 for Injection
- Placebo (Placebo Comparator): (0.9%NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-DUX4 for Injection — single or multiple doses of ARO-DUX4 by intravenous (IV) infusion
  Arms: ARO-DUX4
Drug: Placebo — calculated volume to match active treatment by IV infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of ARO-DUX4 in participants with facioscapulohumeral muscular dystrophy Type 1 (FSHD1). In Part 1 of the study, participants will receive one dose of ARO-DUX4 or placebo. In Part 2 of the study, participants will receive 4 doses of ARO-DUX4 or placebo. Participants who complete Part 1 will have the option to re-screen and re-randomize into Part 2. All participants will undergo pre- and post-dose MRI-guided muscle biopsies (a total of 2 biopsies). Participants who complete Part 1 and enroll in Part 2 will be required to undergo an additional screening biopsy. Participants completing Part 1 or Part 2 may have the option to continue to receive drug in an open-label extension study or may be eligible to participate in later-stage clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed FSHD1 based on Screening evaluation or source verifiable medical record
* Clinical severity score between 3 and 8 (scale, 0 to 10)
* Must have eligible lower extremity muscle for biopsy as determined from MRI by a central reader
* A 12-lead electrocardiogram (ECG) at Screening with no abnormalities that may compromise participant's safety in the study
* Participants of childbearing potential and their partners must use highly effective contraception during the study and for at least 12 weeks following the end of study or last dose of study medication, whichever is later. Males must not donate sperm during the study from Day 1 until at least 12 weeks following the end of study or last dose of study medication, whichever is later.

Exclusion Criteria:

* Human Immunodeficiency Virus (HIV) infection as shown by presence of anti-HIV antibody (seropositive) at Screening
* Seropositive for hepatitis B (HBV) or hepatitis C (HCV) at Screening
* Uncontrolled hypertension
* Severe cardiovascular disease
* History of thrombolic events
* Platelet count less that the lower limit of normal at Screening
* History or presence of: a hypercoagulable state, nephrotic range proteinuria, antiphospholipid antibody syndrome, myeloproliferative disease, inability to ambulate, use of hormone-based contraceptives.
* Any contraindication to muscle biopsy or MRI

Note: additional inclusion/exclusion criteria may apply per protocol

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Over Time Through End of Study (EOS) | Part 1: Up to Day 90; Part 2: Up to Day 360

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARO-DUX4: Maximum Observed Plasma Concentration (Cmax) | Part 1: through 48 hours post-dose (all cohorts) and through 48 hours post second dose (Cohorts 3 & 4 only); Part 2: through 8 hours post first and second dose
PK of ARO-DUX4: Area Under the Plasma Concentration Versus Time Curve from Zero to 24 Hours (AUC0-24) | Part 1: through 48 hours post-dose (all cohorts) and through 48 hours post second dose (Cohorts 3 & 4 only); Part 2: through 8 hours post first and second dose
PK of ARO-DUX4: Area Under the Plasma Concentration Versus Time Curve from Zero to the Last Quantifiable Plasma Concentration (AUClast) | Part 1: through 48 hours post-dose (all cohorts) and through 48 hours post second dose (Cohorts 3 & 4 only); Part 2: through 8 hours post first and second dose
PK of ARO-DUX4: Area Under the Plasma Concentration Versus Time from Zero to Infinity (AUCinf) | Part 1: through 48 hours post-dose (all cohorts) and through 48 hours post second dose (Cohorts 3 & 4 only); Part 2: through 8 hours post first and second dose
PK of ARO-DUX4: Terminal Elimination Half-Life (t1/2) | Part 1: through 48 hours post-dose (all cohorts) and through 48 hours post second dose (Cohorts 3 & 4 only); Part 2: through 8 hours post first and second dose
PK of ARO-DUX4: Systemic Clearance (CL) | Part 1: through 48 hours post-dose (all cohorts) and through 48 hours post second dose (Cohorts 3 & 4 only); Part 2: through 8 hours post first and second dose
PK of ARO-DUX4: Volume of Distribution (Vss) | Part 1: through 48 hours post-dose (all cohorts) and through 48 hours post second dose (Cohorts 3 & 4 only); Part 2: through 8 hours post first and second dose
PK of ARO-DUX4: Recovery of Unchanged Drug in Urine Over 0-24 Hours (Amount Excreted: Ae) | Part 1: through 48 hours post-dose (all cohorts) and through 48 hours post second dose (Cohorts 3 & 4 only); Part 2: through 8 hours post first and second dose
PK of ARO-DUX4: Fraction of Drug Excreted in Urine as Percent of Intravenous (IV) Dose (Fe) | Part 1: through 48 hours post-dose (all cohorts) and through 48 hours post second dose (Cohorts 3 & 4 only); Part 2: through 8 hours post first and second dose
PK of ARO-DUX4: Renal Clearance (CLr) | Part 1: through 48 hours post-dose (all cohorts) and through 48 hours post second dose (Cohorts 3 & 4 only); Part 2: through 8 hours post first and second dose

CONTACTS AND LOCATIONS:
Locations (17):
- Australia (4):
  - Research Site 2, Liverpool, New South Wales
  - Research Site 3, Auchenflower, Queensland
  - Research Site 1, Birtinya, Queensland
  - Research Site 4, Melbourne, Victoria
- Canada (3):
  - Research Site 2, Calgary, Alberta
  - Research Site 3, Edmonton, Alberta
  - Research Site 1, Montreal, Quebec
- Germany (2):
  - Research Site 2, München
  - Research Site 1, Ulm
- Italy (2):
  - Research Site 1, Milan
  - Research Site 2, Roma
- Research Site 1, Leiden, Netherlands
- Research Site 1, Auckland, New Zealand
- Spain (3):
  - Research Site 3, Barcelona
  - Research Site 2, Madrid
  - Research Site 1, Valencia
- Research Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No